CLINICAL TRIAL: NCT05763784
Title: Percutaneous TightRope Fixation for Traumatic Pubic Symphysis Diastasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study plan has halted and was withdrawn from the IRB.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Simon Tiziani, Postdoctoral Trainee, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-1070
Record Dates: First submitted 2022-07-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Pubic Symphysis Diastasis
MeSH Terms: conditions — Pubic Symphysis Diastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pelvic Tightrope fixation (Experimental): Theses patients will be treated with Tightrope for their traumatic pubic symphysis diastasis
  Interventions: Device: Tightrope

INTERVENTIONS:
Device: Tightrope — Tightrope use special fiber and a set of metal buttons to fix diastasis of a joint.

SUMMARY:
This study is done to evaluate the safety of a minimal anterior approach to the pubis symphysis and to examine the efficacy of TightRope for internal fixation of pubic symphysis traumatic diastasis.

DETAILED DESCRIPTION:
Pelvic ring injuries are a challenging task for the orthopaedic surgeon. Commonly, these are associated with hemorrhagic shock, head injury and abdominal trauma. Mortality rate is high and ranges between 11 and 57 percent Pelvic ring injuries are found in polytrauma patients. As such, perioperative complications are not uncommon and comprise shock, sepsis, acute respiratory distress syndrome (ARDS), Multiorgan dysfunction syndrome (MODS), compensatory anti-inflammatory response syndrome (CARS) , sexual dysfunction , and chronic pain.

Reduction and fixation of these injuries is difficult due to complex pelvic anatomy and powerful deforming musculature forces. Often, anatomical restoration requires extensile exposures with considerable biologic burden on the already injured patient. Open reduction is a risk factor for surgical site infections and possible sepsis. The latter is highly associated with increased Body Mass Index (BMI) and risk of postoperative infection.

Minimal invasive pelvic surgery, using closed reduction and percutaneous screws can reduce intraoperative blood loss and shock, decrease mortality rates, postoperative infections and sepsis. In addition, minimal invasive surgery has been shown to be as effective as formal open reduction surgery. Patients with soft tissue compromise such as degloving injuries or burns can also benefit from incorporating minimal invasive surgery.

Internal fixation of pelvic injury is broadly classified to posterior elements (Sacrum, Sacroiliac joint and Sacrotuberous and sacrospinous ligaments) and anterior elements (Pubic symphysis, pectineal ridge and rami). Currently, percutaneous fixation of the Sacroiliac components is widely done, however, formal open reduction using an extensive approach and symphyseal plating remains the gold standard for fixation of the pubis symphysis diastasis.

Currently the management of symphyseal injuries is still one that the overwhelming body of pelvic surgeons would still treat with open reduction and plating via a Pfannenstiel approach. This is because of the relative ease of accessibility to the anterior pelvic ring, good access to the surgical target, low incisional hernia rates and perceived low infection rates. This technique is not without its disadvantages though. The approach requires dissection through a complex anatomical region. Access for plate insertion often requires lateral incision extension, particularly in larger patients. This can increase the risk of damage to inguinal canal and its contents. This can result in ongoing pain symptoms. The approach also sometimes requires the detachment of the distal insertion of the rectus abdomens muscles. The sequelae of this were discussed by Pennal In this study the investigator aims to test a new pubic symphysis diastasis fixation strategy, using the TightRope device combined with a percutaneous anterior approach. TightRope device (Arthrex) is wildly used in orthopaedic surgery for ankle syndesmotic fixation . This device utilizes two metal buttons that can be inserted to attach to bone segments, through a single drill hole. Compression between the two buttons is achieved by pooling the external threads. Following proper reduction and sufficient compression the device is automatically fixed by a locking mechanism in the superficial button. TightRope has been shown to be as strong as conventional 3.5 mm stainless steel screws used in pubic symphysis fixation . In addition, TightRope fixation can potentially decrease the high failure rate of symphyseal plating, reporting to be between 12-33%. In this study a custom-made TightRope prototype made for symphysis diastasis will be used.

The scope of the study is to evaluate the safety of a minimal anterior approach to the pubis symphysis and to examine the efficacy of TightRope for internal fixation of pubic symphysis traumatic diastasis. The authors believe that this fixation method will be more stable then cannulated screws and as stable as plating. In addition, investigator believes that avoiding extensile approach needed for plating will have a positive effect on patient's outcome and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18. Pelvic injury with pubic symphysis diastasis necessitating internal fixation. The study will include both English and Spanish speaking patients.

Exclusion Criteria:

* Age under 18, hemodynamic instability, Pregnancy, concomitant acetabular fracture, malignancy, open fracture. patient not able to understand and sign informed consent (English and Spanish).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Diastasis healing as measured by x-ray. | 2 years
  Diastasis healing will be measured by x-ray. x-ray images will be taken during the initial procedure and on each follow-up. The distance will be measured from the most medial side of each side of the superior rami. Any widening will be compared to post operative x-ray and measured in centimeters. The bigger the gap the less stabilized the pubic symphysis.

IPD SHARING:
Plan to Share IPD: No